CLINICAL TRIAL: NCT01099592
Title: Predictors of Depression Treatment Response Following an Acute Coronary Syndrome
Brief Title: Antidepressants to Promote Recovery of Cardiac Patients Suffering From Depression
Acronym: ARCADE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: inability to recruit
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Nancy Frasure-Smith, Associated Researcher, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 10.004
Record Dates: First submitted 2010-04-01; First posted 2010-04-07 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Acute Coronary Syndrome; Major Depressive Episode
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Citalopram — All patients will take citalopram once daily. Medication will be commercial tablets of 20 mg or 40 mg. All patients will start on a half dose of 10 mg and, if there are no severe side effects, will be increased to 20 mg after 1 week, and if the HAMD-24 at 6 weeks is not < 8, the dose will increase to 40 mg.
  Other Names: celexa

SUMMARY:
Depression is frequently seen in cardiac patients. It has been shown that depression often has a negative impact on the course of coronary disease. More recently, research has demonstrated that some antidepressants can be used safely to treat depressed coronary patients. Although the majority of patients improve substantially with antidepressant treatment, a significant proportion do not respond to antidepressants. This project seeks to better understand why depression does not improve equally well in all patients. Ultimately, the hope is to improve the treatments available to people affected by both cardiac disease and depression, and to help select the best type of treatment in advance for each individual based on his or her personal history, and biological characteristics.

DETAILED DESCRIPTION:
In this study 140 patients who have had a recent hospitalization for an acute coronary syndrome and who have major depression will all receive 12 weeks of treatment with the antidepressant citalopram and regular clinical management visits from a mental health professional. The objective is to examine the characteristics of depressed cardiac patients who do and do not show an improvement in depression with citalopram treatment. There is evidence that the causes of depression may be different in some people with cardiac disease than in individuals who do not have heart problems, and these differences may be at least partially involved in determining response to antidepressant treatment. Inflammation, one of the body's responses to the development of atherosclerosis (hardening of the arteries and blockages in the heart) may be particularly important in producing depression in cardiac patients. There may also be changes in the body's metabolism of tryptophan, a protein that is involved in making serotonin, and levels of serotonin are often low in depression. Other factors thought to influence the development of depression include childhood experiences and personality factors. Heredity and family history also seem to play a role in some people with depression and heart disease. Finally, some patients experience sleep apnea, interruptions in breathing while they are asleep, that can contribute to both cardiac disease and depression.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnostic and Statical Manual-Revision 4 (DSM-IV) diagnosis of current MDD based on the Structured Clinical Interview for Depression (SCID)
* Duration of major depressive disorder (MDD) at least 4 weeks at baseline
* Hospital discharge for an acute coronary syndrome 4 to 24 weeks prior to baseline
* No coronary artery bypass (CABG) surgery during or since the admission for the index event, and no plan for CABG during the next 4 months after baseline
* Stable coronary artery disease (CAD) based on physician's clinical judgement
* Provision of informed consent

Exclusion Criteria

* Significant cognitive problems (Mini-mental Status Exam, MMSE < 24) Structured Clinical Interview for Depression (SCID) documented bipolar disorder or use of lithium or anticonvulsants (e.g. tegretol, depakene, neurontin) for mood disorder
* MINI International Neuropsychiatric Interview (MINI) documented major depression with psychotic features
* MINI documented current or recent (within 12 months) substance abuse or dependence
* Serious suicide risk based on clinical judgment
* Currently taking antidepressants (including St. John's Wort)
* Absence of response to a previous adequate trial of citalopram
* Lifetime evidence of citalopram intolerance or lifetime evidence of intolerance to two or more other SSRIs
* 2 or more previous unsuccessful trials of treatment for the current depressive episode
* Depression due to a general medical condition based on clinical judgment (e.g., clinical hypothyroidism)
* Cold, flu or other infection or dental work (including teeth cleaning) in 14 days before baseline
* Use of antibiotics or steroids (other than topical steroids) in 14 days before baseline
* Participation in any randomized clinical trial
* Inability to speak French or English
* Investigator's judgement that patient is unable/unwilling to comply with study regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to 12 weeks in depression levels on the 24-item Hamilton Depression Rating Scale (HAMD-24) | 12 weeks
  Administered centrally by telephone

SECONDARY OUTCOMES:
Changes from baseline to 12 weeks in depression levels on the Inventory of Depressive Severity Clinician Version (IDS-C) | 12 weeks
  Administered centrally by telephone
Changes from baseline to 12 weeks in self-reported depression symptoms on the Beck Depression Inventory-II (BDI-II) | 12 weeks
  self-report
Changes from baseline to 12 weeks in Inflammatory markers | 12 weeks
  e.g. Tumor necrosis factor-alpha (TNF-alpha), Interleukin-6 (IL-6), Interleukin-10 (IL-10), C-Reactive Protein (CRP), Soluble intercellular adhesion molecule-1 (s-ICAM1)
Changes from baseline to 12 weeks in kynurenine levels | 12 weeks
Changes from baseline to 12 weeks in tryptophan levels | 12 weeks
Changes from baseline to 12 weeks in neopterin levels | 12 weeks
Changes from baseline to 12 weeks in cognitive function | 12 weeks
  scores on the Trail Making Tests A and B, Digit Symbol Substitution Test, Rey Auditory Verbal Learning Test

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Frasure-Smith, PhD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal; François Lespérance, MD, Principal Investigator — Département de psychiatrie, Centre Hospitalier de l'Université de Montréal
Locations (2):
- Canada (2):
  - Centre de recherche du CHUM, Montreal, Quebec
  - Montreal Heart Insitute, Montreal, Quebec